CLINICAL TRIAL: NCT06864650
Title: Effectiveness of Ergonomic Training and Exercise in Automotive Factory Workers With Nonspecific Chronic Low Back Pain: a Randomized Controlled Trial
Brief Title: Effectiveness of Ergonomic Training and Exercise in Automotive Factory Workers With Nonspecific Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar25
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Work-related Illness
MeSH Terms: interventions — Ergonomics; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ergonomics training (Active Comparator): group without any intervention
  Interventions: Other: Ergonomics training
- Ergonomics training +exercise program (Experimental): The group that followed the 12-week exercise program
  Interventions: Other: Ergonomics training; Other: exercise program

INTERVENTIONS:
Other: Ergonomics training — Each of the control group participants will receive separate ergonomics training. The content of this training will include the topics of "what is ergonomics, the purpose of ergonomics, musculoskeletal diseases in employees, work-related musculoskeletal risk factors."
Other: exercise program — stretching exercises strengthening exercises waist exercises core exercises relaxation exercises
  Arms: Ergonomics training +exercise program

SUMMARY:
This study compares the effectiveness of ergonomic training and exercise in automotive factory workers with chronic low back pain of unknown cause.

DETAILED DESCRIPTION:
The study was planned as a randomized controlled study. Workers between the ages of 18-60 who have back pain and work in an automotive factory in Galway, Ireland will be included in the study. Participants will be divided into two groups. The factory workers included in the study will be divided into a study group and a control group using a simple random method. Randomization will be done using the sealed envelope method. The study group will be given stretching and strengthening exercises along with ergonomics training. The control group will be given only ergonomics training. The exercises they will do and the ergonomics training will be explained to the participants individually and supported with a brochure. The participants will be asked to do the given exercises 3 days a week and continue for 12 weeks. The given exercises will be followed up with an exercise follow-up chart. In order to collect data on the sociodemographic characteristics of the participants, a personal information form will be prepared by the researcher and the participants will be asked to fill it out. In order to collect data from the participants; Visual Analog Scale will be used to collect information about pain, International Physical Activity Questionnaire to collect information about physical activity levels, Pittsburgh Sleep Quality Questionnaire to determine sleep quality, Oswestry Low Back Pain Scale for functionality assessment, Manual Muscle Testing to determine muscle strength. These questionnaires will be repeated before starting the study and at the end of the study. The data to be obtained will be evaluated using SPSS 24 package program.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-60 years old
* Having worked in the same factory for at least 2 years
* Working full time
* Having complained of back pain for at least 3 months
* visual analog scale>4, pain 4 and above on visual analog scale

Exclusion Criteria

* Being under 18 years old or over 60 years old
* Having worked for less than 2 years
* Working part time
* Having complained of back pain for less than 3 months
* visual analog scale Presence of psychological problems
* Using sleeping pills
* Having undergone surgical intervention in the last 6 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
Oswestry Low Back Pain Disability Questionnaire | 14 weeks
  It was developed to measure the functionality of individuals. The scale determines functional disability for activities such as sitting, walking, personal care, lifting, social life, travel, and sleep. There are 10 questions in this scale. Each question has 6 options. Participants are asked to choose the definition that best describes their situation from these options. A score of 0-5 is assigned for each of the sentences, and the highest possible score is 50 points. It is evaluated as mild between 1 and 10 points, moderate between 11 and 30 points, and severe between 31 and 50 points.
The Pittsburgh Sleep Quality Index | 14 weeks
  Pittsburgh Sleep Quality Index; It evaluates sleep duration, sleep disturbance, sleep efficiency, subjective sleep quality, sleep medication use, daytime dysfunction, and sleep delay and consists of a total of 24 questions. 19 of them are self-report scales and 5 of them consist of questions to be answered by a friend or spouse. There are 7 components with 18 questions scored in the scale, and each component is evaluated between 0 and 3 points. The total score ranges from 0 to 21, and 5 or more is an indicator of "poor sleep quality
Short form of the International Physical Activity Questionnaire | 14 weeks
  It consists of 8 questions with a recall period defined as 'last week'. The questions of the scale ask whether the participant walks for at least 10 minutes on any given day or does moderate or vigorous activities, and how much time/day the individual spends on each of these activities.

CONTACTS AND LOCATIONS:
Overall Officials: Kübra TOSYALI, Study Chair — Uskudar University
Locations (1):
- Valeo Vision System, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stieglitz DD, Vinson DR, Hampton MC. Equipment-based Pilates reduces work-related chronic low back pain and disability: A pilot study. J Bodyw Mov Ther. 2016 Jan;20(1):74-82. doi: 10.1016/j.jbmt.2015.06.006. Epub 2015 Jun 15. PMID 26891640
- [Background] Chenot JF, Greitemann B, Kladny B, Petzke F, Pfingsten M, Schorr SG. Non-Specific Low Back Pain. Dtsch Arztebl Int. 2017 Dec 25;114(51-52):883-890. doi: 10.3238/arztebl.2017.0883. PMID 29321099
- [Background] Pehlevan E, Sevgin O. Effect of exercise given to factory workers with ergonomics training on pain and functionality: A randomized controlled trial. Work. 2024;78(1):195-205. doi: 10.3233/WOR-230663. PMID 38701125